CLINICAL TRIAL: NCT04346953
Title: Investigation Of The Effectiveness Of Video-Based Exercise Program Applied To Adult Individuals Who Experience Social Isolation At Houses Due To The Coronavirus (COVID-19) Pandemic
Brief Title: Video-Based Exercise for Individuals With Social Isolation Due to Coronavirus (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Healthy Lifestyle
Keywords: Social isolation; Exercises; Physical inactivity; Health benefits
MeSH Terms: conditions — Social Isolation; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group to which the exercise videos consisting of aerobic and strengthening exercises will be applied.
  Interventions: Behavioral: Video based exercise
- Control Group (No Intervention): The control group where only the evaluations will be made and information about the benefits of exercise will be given.

INTERVENTIONS:
Behavioral: Video based exercise — Individuals (n = 64) to be included in the study group will be grouped according to the levels of physical activity (low, medium, high level) determined by the International Physical Activity Questionnaire. An exercise program will be created for each group based on physical activity levels and videos of these exercise programs will be prepared. The videos will be scheduled for 20 minutes. Individuals will be asked to apply for these programs with video for 20 minutes every day for 6 weeks. Exercise programs will start with pulmonary exercises and warm-up exercises to prepare for exercise. The exercise program will end with cool down exercises. The exercise protocol will be determined as a combination of aerobic and strengthening exercises.
  Arms: Study Group

SUMMARY:
In December 2019, new coronavirus pneumonia (COVID-19) broke out in Wuhan (Hubei, China), and it spread rapidly from one city to the whole country in just 30 days, and then worldwide cases began to appear. All the countries of the world take some precautions to prevent the spread of this epidemic disease, which WHO declared as "pandemic". Apart from compulsory situations, non-home and social isolation are the primary measures. However, not leaving the house and social isolation brings with it the restriction of physical activity.

According to World Health Organization (WHO), in order to obtain health benefits, adult individuals between the ages of 18-64 should perform at least 150 minutes of physical activity per week (30 minutes a day for 5 days a week) or intensive physical activity for at least 75 minutes a week. For additional health benefits, adults should increase their moderate-intensity physical activities to at least 300 minutes a week or equivalent. Physical activity; It is directly related to the prevention of chronic diseases, increasing fitness, strengthening the muscles and increasing the quality of life. It is reported that one of the ten main risk factors in terms of mortality in the world is insufficient physical activity. The effects of social isolation are related to physical inactivity, smoking and the possibility of having both health risk behaviors together. Practical and innovative interventions are needed to reduce physical performance and decrease in muscle mass, strength and physical performance in the aging population. Considering today's conditions and current COVID-19 Pandemic, technology-supported exercise programs are effective in increasing the motivation for physical activity. The purpose of this study; In order to prevent the spread of the COVID-19 pandemic, social isolation, which is one of the measures taken in our country, is to evaluate the physical activity level of adults and to investigate the effectiveness of home exercises. It is aimed to use a model based on the video supported by a home-based exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-60 years old
* Being in social isolation due to COVID-19 virus
* Not having any physical disability that prevents them from doing physical activities
* Being in social isolation due to COVID-19 virus
* Having access to exercise videos

Exclusion Criteria:

* Having a serious cognitive impairment
* Having serious hearing and vision problems
* Having vestibular disorders that can cause loss of balance
* Having diabetes and/or hypertension or a neurological disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | 2 weeks
  The International Physical Activity Questionnaire -Short Form (IPAQ-SF) measures the frequency and duration of moderate physical activity, vigorous physical activity, walking, and sedentary behavior using 7 questions and is considered more suitable for population surveillance and large-scale studies compared with the long form . The IPAQ-SF was validated for adults.According to the score obtained, the physical activity levels of individuals are determined. It indicates lower physical activity level below 600 Metabolic Equivalent Threshold (MET)-min per week, medium physical activity level between 600-3000 Metabolic Equivalent Threshold (MET)-min per week and high physical activity level between 600-3000 Metabolic Equivalent Threshold (MET)-min per week.
Nottingham Health Profile | 2 weeks
  Nottingham Health Profile was created in England in 1985 to evaluate the quality of life-related to health. The Nottingham Health Profile is a general quality of life questionnaire that assesses the level of individuals health problems and how they affect their daily life activities.
Beck Depression Inventory | 2 weeks.
  It is among the most used scales to measure depression all over the world. It consists of 21 questions in total. Each item gets points between 0-3. 11-17 points indicate mild depression, 18-29 points indicate moderate depression, and 30-63 points indicate severe depression.
Beck Anxiety Inventory | 2 weeks
  It is used to evaluate the anxiety symptoms experienced by individuals due to social isolation. It consists of 21 items and is scored between 0-3. It indicates low anxiety of 0-21 points, moderate anxiety of 22-35 points and high anxiety of 36 points and above.
Pittsburgh Sleep Quality Index | 2 weeks
  It is a scale that provides information about sleep quality and type and severity of sleep disorder in the last month. The sleep quality of the person on this scale; sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use and daytime dysfunction. Each question is given a score of 0-3. High scores reflect poor sleep quality. If the total score obtained from the scale is less than 5, it is defined as "Good sleep quality" and 5 and above is defined as "Bad sleep quality".
Timed Get Up and Go Test | 2 weeks
  Used for mobility assessment. The test begins while the person is sitting in the chair. The person is asked to get up from the chair, walk 3 meters, come back and sit on the chair again, and the time is recorded. If an elderly person completes the test for more than 12 seconds, there is a risk of falling.
Flamingo Balance Test | 2 weeks
  Flamingo Balance Test will be used to evaluate the static balance of the individuals who will participate in the study. This test is done on one foot. While individuals are in balance with one foot, time begins and tries to stay in balance for 1 minute. The time is stopped when the balance is disturbed. When the time is completed, each individual attempt to balance is counted and this number is recorded as the individual's score at the end of the test. If the individual tries to balance 15 times in the first 30 seconds, the test is stopped and zero points are given.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)